CLINICAL TRIAL: NCT02213822
Title: MOLECULAR TESTING OF CANCER BY INTEGRATED GENOMIC, TRANSCRIPTOMIC, AND PROTEOMIC ANALYSIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2055-13
Record Dates: First submitted 2014-07-31; First posted 2014-08-12 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-07

CONDITIONS: Solid Tumors; Hematological Malignancies
Keywords: genome; transcriptome; molecular; proteome; oncogenic mutations; sequencing; solid tumor; hematological malignancy; cancer; analysis; genetic; mutation
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tissue, blood, saliva, body fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pts with Solid Tumors/ Hematological Cancer: Patients on this study must have either a suspected or confirmed solid tumor or hematological cancer. The intervention performed in this study is the molecular analysis of cancer. The samples will be taken at the time of the patient's planned diagnostic or staging procedure. If the patient is scheduled for surgery a sample of tissue not required for their diagnosis will be obtained and used for this research study. If the patient has undergone a previous diagnostic procedure, some of the stored tissue from that procedure will be submitted for molecular analysis as well.
  Interventions: Other: Molecular Analysis of Cancer

INTERVENTIONS:
Other: Molecular Analysis of Cancer — The intervention performed in this study is the molecular analysis of cancer. Samples to be tested for genetic alterations will be collected during the course of a routine diagnostic procedure such as a surgery or tumor biopsy. Samples that have been stored from previous diagnostic procedures will be analyzed as well. This testing will be performed by the Department of Pathology at Rhode Island Hospital or an outside laboratory designated by Rhode Island Hospital. The extent of molecular testing will be different in each individual case. For example, in some cases, study of genetic alterations will start with whole genome or exome sequencing and will be confirmed by targeted Sanger resequencing, single nucleotide polymorphism, and transcriptome analysis. In other cases targeted multigene panel sequencing or targeted amplicon Sanger sequencing will be the initial and only step.

SUMMARY:
The purpose of this study is to discover genetic changes associated with different cancers. With the information from this study the investigators hope to provide better ways to prevent, detect and treat many cancers.

Many diseases can result from changes in a person's genetic material that causes cells to not work properly. Currently, researchers and doctors know some of the genetic changes that can cause disease, but they do not know all of the genetic changes that can cause disease.

This project is designed to identify genetic changes that can cause cancer in humans. Specimens will be collected from a scheduled diagnostic or routine (i.e. blood draw for counts) procedure and may include samples from the tissue itself (surgery), bone marrow, blood, saliva, urine, spinal fluid, sputum, joint fluid, seminal fluid, ascites (a fluid that fills up in the abdomen), and/or pleural fluid (fluid in the lung cavity), to either confirm the diagnosis of cancer or to help to decide how best to treat cancer or other illness. Additionally archived tissue may be analyzed. Samples may be stored for future use in later experiments. The Department of Pathology at Rhode Island Hospital will store the samples.

Information from the medical record, such as responses to treatments or family history of cancer, will be collected.

DETAILED DESCRIPTION:
Complex, progressive, multigenic, somatic mutations of the genome are now widely accepted as the primary driving force in the evolution of cancer initiation, growth, metastasis and pharmacoresistance. Different types of tumors are associated with mutations in distinct sets of genes, and there is a pressing need for a sequencing-based method of analyzing panels of candidate genes that differ for each tumor type.

Traditional approaches to sequence analysis employing capillary electrophoresis-based Sanger sequencing are widely used to guide therapy for patients with lung and colorectal cancer and for melanoma, sarcomas, leukemias and lymphomas. This technology is limited in throughput, scalability, speed, and resolution. The emerging technology such as next-generation sequencing (NGS) - holds a number of advantages over traditional methods, including the ability to fully sequence large numbers of genes in a single test and simultaneously detect deletions, insertions, copy number alterations, translocations, and exome-wide base substitutions in all known cancer-related genes.

Sequencing the whole genome is financially prohibitive for many potentially valuable applications. One alternative to whole genome methods is target enrichment, such as exome sequencing, which captures and sequences only protein coding regions. The exome represents 1-2% of the human genome; however contains the vast majority of disease causing alterations. In addition to exome sequencing, full-length transcriptome (mRNA) sequencing offers a fast and inexpensive alternative. It is an easier method to identify coding sequences and capture variants in genes that are expressed, as well as to generate additional information, such as gene expression level and splicing patterns.

The goal of this study is to investigate genomic, transcriptomic and proteomic alterations in human solid cancers and hematologic malignancies.

Patients >18 y.o. diagnosed with cancer (including any solid tumor or hematologic malignancy) or patients who are undergoing a procedure for the diagnosis of a presumed cancer are eligible.

The research analysis will be performed by the department of pathology or the division of hematology oncology. The body/blood tissue analyzed will be from extra tissue/blood that is not needed for diagnosis or evaluation of the patient's cancer. All samples will be de-identified. Samples will be stored for an indefinite period of time or until all samples are utilized.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent
* Patient has either a suspected or confirmed solid tumor or hematological malignancy
* There is enough tissue or body fluid to allow for experimental study
* The patient is over the age of 18

Exclusion Criteria:

* The patient is unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in this study will have either a suspected or confirmed solid tumor or hematological malignancy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The Frequency of "Actionable" Oncogenic Mutations | 1 year
The Prevalence of Genomic, Transcriptomic, and Proteomic Abnormalities in Human Cancer | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Perez, M.D., Principal Investigator — Lifespan Corporation
Locations (3):
- United States (3):
  - Rhode Island Comprehensive Cancer Center at East Greenwich, East Greenwich, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island